CLINICAL TRIAL: NCT04051138
Title: The Effect of VOXX/eSmartr High Performance Technology on Sports Vision Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChampionsEdge, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Voxx1
Record Dates: First submitted 2019-08-05; First posted 2019-08-09 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Vision, Binocular; Sports Medicine

STUDY DESIGN:
Intervention Model Description: randomized, double blind, prospective
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Voxx socks and sleeves — participants will be tested with a true device as well as with a placebo device

SUMMARY:
This study is designed to compare the effect of Voxx/eSmartr technology on common measures of sports vision performance including (Hand-Eye Coordination/Reaction time, visual concentration and basic visual functions of size detection and contrast sensitivity). The study will be a randomized, prospective, double-blind design in order to determine the effect of this technology on a subject's sports vision ability.

ELIGIBILITY:
Inclusion Criteria.

* Female or Male age 18-45 years of age
* Exercises at least once a week by self-report
* Physically able to complete the HEC/RT test (e.g. no shoulder or arm discomfort or limitation

Exclusion Criteria.

* Member of a vulnerable population
* Visual or physical condition which precludes performing the physical or visual testing (e.g. strabismus, double vision, shoulder or arm pain or injury)
* Previous training in hand-eye coordination/reaction time or visual concentration
* History of double vision or strabismus
* Insufficient vision to drive an automobile in NY State

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
CoreScore | 1 day
  A measure of visual function scored on a linear scale fro +5 to -5, more positive scores are better

SECONDARY OUTCOMES:
Hand-Eye Coordination/Reaction Time | 1 day
  A measure of how fast the subject reacts to a visual target with their hand, scored on milliseconds, faster the better
Neurotracker score | 1 day
  A measure of how correctly the subject can track multiple objects, scored from 0 to 5 with higher score being better

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Laby, MD, Principal Investigator — ChampionsEdge, LLC
Locations (1):
- SportsVisionNYC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No